CLINICAL TRIAL: NCT04381754
Title: Use of Implanting the Biotronik Passeo-18 Lux Drug Coated Balloon to Treat Failing Hemodialysis Arteriovenous Fistulas and Grafts
Brief Title: Use of Implanting the Biotronik Passeo-18 Lux Drug Coated Balloon to Treat Failing Haemodialysis Arteriovenous Fistulas and Grafts.
Acronym: SEMPER FI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1.5
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Arterio-venous Fistula; Dialysis Access Malfunction; Hemodialysis Access Failure; Arteriovenous Graft Stenosis
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AVG/AVF Treated with Passeo-18 Lux: Patients with failing dialysis access, treated lesions located between the anastomosis to the axillary-subclavian vein junction.
  Interventions: Device: Passeo-18 Lux

INTERVENTIONS:
Device: Passeo-18 Lux — Patients with significant inflow or outflow stenosis between the anastomosis to the axillary-subclavian vein junction, as defined by the insertion of the cephalic vein, who had undergone fistuloplasty with Passeo-18 Lux
  Other Names: Biotronik

SUMMARY:
The most common problem with haemodialysis arteriovenous fistulas (AVF) and arterio-venous grafts (AVG) is stenosis, which can lead to inadequate dialysis, and eventual access thrombosis. Conventional plain old balloon angioplasty is associate with high recurrence rates of stenosis and repeated interventions. The advent of successful drug-eluting technology in the treatment of the coronary vascular bed and subsequent positive accumulating evidence in the peripheral arterial circulation has prompted the use of drug coated balloons (DCB) in the access fistula circuit for venous stenosis and in-stent restenosis. Recent studies suggest that DCBs may significantly reduce re-intervention rates on native and recurrent lesions. The restenosis process is in part or in whole the result of neo-intimal hyperplasia (NIH) and NIH is considered the main culprit in access circuit target lesion stenosis. NIH is the blood vessel's healing response to the barotrauma from the angioplasty process. A critical component of NIH is the cellular proliferative stage with mononuclear leucocytes identified as the primary inflammatory cell type involved. The rationale for drug elution is to block the NIH response with an anti-metabolite such as paclitaxel. It is important to emphasize that the role of drug elution in the treatment of vascular stenosis is not to obtain a good haemodynamic and luminal result but to preserve a good result obtained during POBA from later restenosis due to NIH and minimise reinterventions and readmissions to hospital for what is a frail population of patients.

A meta-analysis performed by Khawaja et al. seemed to suggest that DCBs conferred some benefit in terms of improving target lesion primary patency (TLPP) in AVFs. An updated meta-analysis performed by our own institution recently showed that DCB appears to be a better and safe alternative to conventional balloon angioplasty (CBA) in treating patients with HD stenosis based on 6- and 12-months primary patency and increased intervention free period.

The Passeo-18 Lux (Biotronik Asia Pacific Pte Ltd (Singapore)) drug-coated balloon (DCB) is packaged with a low dose of paclitaxel. Recent studies have shown that low dose coating of paclitaxel with this DCB is useful for preventing restenosis, decrease lumen loss and target lesion revascularization in the peripheral vasculature6 but has not been tested in the dialysis access circuit.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥21 years and ≤90 years
* Native AVF was created more than 2 months prior to the index procedure and had undergone 10 or more hemodialysis sessions utilizing 2 needles
* Target lesion location had to be located between the anastomosis to the axillary-subclavian vein junction, as defined by insertion of the cephalic vein.
* On initial fistulogram, target lesion stenosis had to be >50% on angiographic assessment and in keeping with the clinical indicator for intervention
* Stenosis had to be < 10cm in length to allow for potential treatment with one PCB (length 12 cm) only
* Stenosis had to be initially treated successfully with a high-pressure plain balloon prior to PCB treatment as defined by:

  1. No clinically significant dissection
  2. No extravasation requiring treatment/stenting
  3. Residual stenosis ≤20% by angiographic measurement
  4. Ability to completely efface the lesion waist using the pre-dilation balloon
* No more than one additional ("nontarget") lesions in the access circuit that had to be also successfully treated (≤30% residual stenosis) before drug elution. Separate lesion was defined by at least 3 cm in distance from the target lesion.
* Reference vessel diameter 4mm - 8mm

Exclusion Criteria:

* Women who were pregnant, lactating, or planning on becoming pregnant during the study
* Subject had more than two lesions in the access circuit
* Subject had a secondary non-target lesion that could not be successfully treated
* Sepsis or active infection
* Asymptomatic target lesions
* A thrombosed access or an access with thrombosis treated ≤30 days prior to the index procedure
* Surgical revision of the access site performed, planned or expected ≤ 3 months before or after the index procedure
* Patients who were taking immunosuppressive therapy or are routinely taking ≥ 15 mg of prednisone per day;
* Currently participating in an another investigational drug, biologic, or device study involving sirolimus or paclitaxel
* Contraindication to aspirin or clopidogrel usage
* Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, or language barrier such that the subject is unable to give informed consent
* Uncooperative attitude or potential for non-compliance with the requirements of the protocol making study participation impractical
* Where final angioplasty treatment requires a stent or drug eluting balloon > 8mm in diameter
* Metastatic cancer or terminal medical condition
* Blood coagulation disorders
* Limited life expectancy (< 12 months)
* Allergy or other known contraindication to iodinated media contrast, heparin or paclitaxel

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a native upper limb AVF or AVG, that is currently in use for haemodialysis, which has a significant inflow or outflow stenosis. Significant stenosis defined as diameter greater than 50% compared to adjacent normal segment and/or other evidence of AVF malfunction. Malfunction defined as the AVF performing inadequate dialysis and clinical signs of a failing dialysis access. Inadequate fistula volume flow - Qa as measured by ultrasound < 500mL/min as probably inadequate. Dialysis numbers: - Qb - a significant stenosis is suggested when the pump speed is < 200ml/min, venous pressure is > 140 mmHg and/or arterial pressure > - 100mmHg. Maximum of 2 discrete stenoses (separated by > 3cm) are allowed to be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
6-month Target Lesion Primary Patency | 6-month post-procedure
  Patency with no re-intervention to the area 5mm proximal to, within, and 5mm distal to, the index treatment segment. TLPP ends when any of the following occur: 1) clinically driven re-intervention to the treatment segment 2) thrombotic occlusions that includes the treatment segment 3) surgical intervention that excludes the treatment segment from the access circuit 4) abandonment of the AVF/AVG due to an inability to treat the treatment segment

SECONDARY OUTCOMES:
Primary Patency | 12 months post-op
  A duration of time measuring intra-access patency that starts from the date of angioplasty with Passeo-18 Lux DCB to the date of one of the following events: thrombosis, or any intervention to facilitate, maintain or re-establish patency (e.g. angioplasty)
Primary assisted patency | 12 months post-op
  Interval date of angioplasty with Passeo-18 Lux DCB until thrombosis
Secondary Patency | 12 months post-op
  A duration of time measuring intra-access patency that starts from the date of angioplasty with Passeo-18 Lux DCB to the date of vascular access abandonment
Number of reinterventions | 12 months post-op
Adverse Events | 12 months post-op
  Intraoperative/perioperative complications, infections, revision surgeries required

CONTACTS AND LOCATIONS:
Overall Officials: Tang Tjun Yip, Principal Investigator — Sinapore General Hospital; Yap Hao Yun, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Troisi N, Frosini P, Somma C, Romano E, Guidotti A, Dattolo PC, Ferro G, Chisci E, Michelagnoli S. Drug-coated balloons reduce the risk of recurrent restenosis in arteriovenous fistulas and prosthetic grafts for hemodialysis. Int Angiol. 2018 Feb;37(1):59-63. doi: 10.23736/S0392-9590.17.03886-X. Epub 2017 Nov 10. PMID 29125264
- [Background] Liao MT, Chen MK, Hsieh MY, Yeh NL, Chien KL, Lin CC, Wu CC, Chie WC. Drug-coated balloon versus conventional balloon angioplasty of hemodialysis arteriovenous fistula or graft: A systematic review and meta-analysis of randomized controlled trials. PLoS One. 2020 Apr 14;15(4):e0231463. doi: 10.1371/journal.pone.0231463. eCollection 2020. PMID 32287283
- [Background] Kennedy SA, Mafeld S, Baerlocher MO, Jaberi A, Rajan DK. Drug-Coated Balloon Angioplasty in Hemodialysis Circuits: A Systematic Review and Meta-Analysis. J Vasc Interv Radiol. 2019 Apr;30(4):483-494.e1. doi: 10.1016/j.jvir.2019.01.012. Epub 2019 Mar 8. PMID 30857987
- [Background] Khawaja AZ, Cassidy DB, Al Shakarchi J, McGrogan DG, Inston NG, Jones RG. Systematic review of drug eluting balloon angioplasty for arteriovenous haemodialysis access stenosis. J Vasc Access. 2016 Mar-Apr;17(2):103-10. doi: 10.5301/jva.5000508. Epub 2016 Feb 5. PMID 26847736
- [Background] Yan Wee IJ, Yap HY, Hsien Ts'ung LT, Lee Qingwei S, Tan CS, Tang TY, Chong TT. A systematic review and meta-analysis of drug-coated balloon versus conventional balloon angioplasty for dialysis access stenosis. J Vasc Surg. 2019 Sep;70(3):970-979.e3. doi: 10.1016/j.jvs.2019.01.082. PMID 31445651
- [Background] Brodmann M, Zeller T, Christensen J, Binkert C, Spak L, Schroder H, Righini P, Nano G, Tepe G. Real-world experience with a Paclitaxel-Coated Balloon for the treatment of atherosclerotic infrainguinal arteries: 12-month interim results of the BIOLUX P-III registry first year of enrolment. J Vasc Bras. 2017 Oct-Dec;16(4):276-284. doi: 10.1590/1677-5449.007317. PMID 29930661